CLINICAL TRIAL: NCT00066859
Title: A Phase III Double-Blind Randomized Trial Comparing Sertraline (Zoloft) And Hypericum Perforatum (St. John's Wort) In Cancer Patients With Mild To Moderate Depression
Brief Title: Sertraline Compared With Hypericum Perforatum (St.John's Wort) in Treating Depression
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: REBACCCWFU-98101; U10CA081851 (NIH)
Record Dates: First submitted 2003-08-06; First posted 2003-08-07 (Estimated); Last update posted 2021-09-09 (Actual); Status verified 2021-09

CONDITIONS: Depression; Unspecified Adult Solid Tumor, Protocol Specific
Keywords: depression; unspecified adult solid tumor, protocol specific
MeSH Terms: conditions — Depression | interventions — Sertraline; Hypericum extract LI 160

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm 1: Sertraline (Zoloft) 50 mg (Active Comparator): Zoloft 50 mg by mouth daily for 1 week if tolerated dose may be increased to 100 mg daily for 4 months
  Interventions: Drug: Zoloft 50 mg
- Arm 2 - St. John's Wort 600mg (Active Comparator): St. John's wort 600 mg daily for 1 week. If tolerated dose may be increased to 900 mg daily for four months.
  Interventions: Dietary Supplement: St. John's Wort 600 mg

INTERVENTIONS:
Drug: Zoloft 50 mg — Zoloft 50 mg by mouth daily for 1 week if tolerated dose may be increased to 100 mg daily for 4 months
  Other Names: Sertraline; Zoloft
  Arms: Arm 1: Sertraline (Zoloft) 50 mg
Dietary Supplement: St. John's Wort 600 mg — St. John's wort 600 mg daily for 1 week, if tolerated. Dose may be increased to 900 mg daily for 4 months.
  Other Names: Hypericum perforatum
  Arms: Arm 2 - St. John's Wort 600mg

SUMMARY:
RATIONALE: Antidepressants such as sertraline and the herb hypericum perforatum (St. John's wort) may be effective in treating mild to moderate depression. It is not yet known which treatment is more effective in improving depression in patients who have cancer.

PURPOSE: This randomized phase III trial is studying how well sertraline works compared to St. John's wort in treating mild to moderate depression in patients with solid tumors.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the change in depression severity in cancer patients with mild to moderate depression treated with sertraline vs Hypericum perforatum.
* Compare the severity of somnolence, nausea, and insomnia in patients treated with these regimens.
* Compare the impact of these regimens on fatigue in these patients.
* Correlate hyperforin concentrations with change in depression severity in patients treated with Hypericum perforatum.

OUTLINE: This is a randomized, double-blind study. Patients are stratified according to level of depression (mild vs moderate), concurrent radiotherapy (yes vs no), and TNM stage (I, II, or III vs IV). Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive oral sertraline daily.
* Arm II: Patients receive oral Hypericum perforatum daily. In both arms, treatment continues for 4 months in the absence of unacceptable toxicity.

Measurements of depression, somnolence, nausea, insomnia, fatigue, and hyperforin concentration are assessed at baseline, and at 1, 2, and 4 months.

PROJECTED ACCRUAL: A maximum of 250 patients will be accrued for this study.

ELIGIBILITY:
INCLUSION CRITERIA:

* Mild or moderate depression as determined by the following criteria (see Section 7.1 and 8.0)
* Mild : HRSD score 10-14; moderate: HRSD score 15-19 (Appendix IV)
* At least 2 of nine symptoms of depression on the PHQ (Appendix V)
* At least one of the nine PHQ symptoms must be either depressed/irritable mood or anhedonia
* Histologically or cytologically documented solid tumor, lymphoma, or primary or metastatic brain tumor > 6 months from radiation with stable disease or no evidence of disease.
* Concurrent cancer chemotherapy with sertraline or St. John's wort is not allowed, therefore patients must have no plan for chemotherapy for 4 months
* Prior chemotherapy is allowed, but patients must be >4 weeks from prior chemotherapy except >6 weeks from prior mitomycin-C or nitrosourea
* Patients receiving Rituxin, Herceptin, Erbitux, Interferon, etc. are eligibile for this study while under treatment.
* Prior or concurrent radiation is allowed except brain irradiation for brain metastases or primary brain tumor. Must be > 6 months from radiation with stable disease or no evidence of disease.
* Age > 18 years
* ECOG performance status 0 -1 (Appendix III)
* Life expectancy >4 months
* Required initial laboratory values (within 3 days of registration): hemoglobin >10 g/dl and bilirubin <1.5 mg/dl, negative pregnancy test
* Signed protocol specific informed consent prior to registration
* Patient recruitment this study will be done through the out patient clinic. The research PI or designee including clinic physician, resident, research nurse or research assistant will review medical information to determine or verify protocol eligibility either at the time the patient is being seen in the clinic for a routine visit/consult or prior to the patient's clinic visit.

EXCLUSION CRITERIA:

* A patient will be excluded if he/she is (a) judged to be severely depressed using the following criteria: HRSD score 20 or more or a positive score on PHQ item i (suicidal ideation) or (b) judged not to be depressed by a score of 9 or less on the HRSD or fewer than two PHQ items scored positively. A patient who is found to be severely depressed or suicidal, either on initial screening or during the trial will be referred for appropriate treatment.
* Psychotic symptoms, dementia, marked agitation requiring medication
* Current or previous alcohol or drug dependence
* Hematologic malignancy (i.e., leukemias, multiple myeloma)
* Planned chemotherapy in the next 4 months
* Antidepressant or St. John's wort use in the last 4 weeks
* Current or planned use of erythropoietin (Procrit®, Aranesp®)
* Current or planned use of theophylline, warfarin (except for central line prophylaxis), protease inhibitors used to treat AIDS, digoxin, cyclosporin, benzodiazepines (such as diazepam, alprazolam, etc), calcium-channel blockers (such as diltiazem, nifedipine, etc), coenzyme A reductase inhibitors (cholesterol lowering agents), macrolide antibiotics (such as azithromycin, erythromycin, clarithromycin, etc), griseofulvin, phenobarbital, phenytoin, rifampin, rifabutin, ketoconazole, fluconazole, itraconazole, corticosteroids, grapefruit juice, or other naturopathic/herbal products that could interfere with St. John's wort (call study chairman with questions).
* Pregnant or nursing women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2004-03-01; Primary Completion 2005-04-01 (Actual); Study Completion 2005-11-01 (Actual)

PRIMARY OUTCOMES:
Depression severity as measured by Hamilton Depression rating scale. | 4 months
  To compare the change in depression severity in cancer patients with mild to moderate depression on sertraline and St. John's wort.

SECONDARY OUTCOMES:
Somnolence, nausea, and insomnia as assessed by the NCI Common Toxicity Criteria. The Epworth Sleepiness Scale will also be used to assess somnolence. | 4 months
Fatigue as measured by the Functional Assessment of Chronic Illness Therapy-Fatigue Scale. | 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Antonius A. Miller, MD, Principal Investigator — Wake Forest University Health Sciences; Edward G. Shaw, MD, Study Chair — Wake Forest University Health Sciences
Locations (6):
- United States (6):
  - Bay Area Tumor Institute, Oakland, California
  - Regional Radiation Oncology Center at Rome, Rome, Georgia
  - CCOP - Central Illinois, Decatur, Illinois
  - CCOP - Southeast Cancer Control Consortium, Goldsboro, North Carolina
  - High Point Regional Hospital, High Point, North Carolina
  - Comprehensive Cancer Center at Wake Forest University, Winston-Salem, North Carolina

IPD SHARING:
Plan to Share IPD: No